CLINICAL TRIAL: NCT01834014
Title: An Exploratory Study to Evaluate Biomarkers as Predictive and /or Prognostic Factors of Benefit From Randomized Phase ll Study of mFOLFOX6+Bevacizumab or mFOLFOX6+Cetuximab in Liver Only Metastasis From KRAS Wild Type Colorectal Cancer
Brief Title: Exploratory Study in Achievement of Improved Survival by Molecular Targeted Chemotherapy and Liver Resection for Not Optimally Resectable Colorectal Liver Metastases
Acronym: ATOM ES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EPS Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOM Exploratory study; UMIN000010429 (Other: UMIN)
Record Dates: First submitted 2013-04-14; First posted 2013-04-17 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Liver Metastasis; Colorectal Cancer
Keywords: Liver only metastasis from KRAS Exon 2 wild type; Liver only metastasis from RAS wild type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFOX + Bmab (Experimental): mFOLFOX plus bevacizumab
  Interventions: Drug: Bevacizumab; Drug: L-OHP; Drug: l-LV; Drug: 5-FU
- mFOLFOX + Cmab (Active Comparator): mFOLFOX plus cetuximab
  Interventions: Drug: Cetuximab; Drug: L-OHP; Drug: l-LV; Drug: 5-FU

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg intravenously administered over 90 minutes (can be reduced to 30 minutes at the minimum) on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Avastin
  Arms: mFOLFOX + Bmab
Drug: Cetuximab — 250 mg/m2 intravenously administered over 60 minutes (400 mg/m2 over 120 minutes as the initial dose) on day 1 and day 8 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Erbitux
  Arms: mFOLFOX + Cmab
Drug: L-OHP — 85 mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Oxaliplatin
Drug: l-LV — 200 mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Levofolinate
Drug: 5-FU — 400 mg/m2 intravenous bolus on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Fluorouracil
Drug: 5-FU — 2400 mg/m2 continuous infusion over 46 hours on day 1 and 2 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Fluorouracil

SUMMARY:
The correlation between the values of angiogenesis-related growth factors in plasma and efficacy, and biomarkers relevant as prognostic factors or predictive factors for sensitivity or resistance to treatment will be examined exploratively.

DETAILED DESCRIPTION:
The correlation between the values of angiogenesis-related growth factors in plasma and efficacy, and biomarkers relevant as prognostic factors or predictive factors for sensitivity or resistance to treatment will be examined exploratively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who registered the ATOM trial and signed informed consent prior to initiation of any trial-specific procedure and treatment.

Exclusion Criteria:

* None

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the values of angiogenesis-related growth factors in plasma with Progression-free survival (PFS) | Baseline, Cycle 8, Progression Disease
  To evaluate the values of angiogenesis-related growth factors in plasma with PFS centrally assessed

SECONDARY OUTCOMES:
To evaluate the correlation of values of angiogenesis-related growth factors in plasma with efficacy and adverse events | Baseline, Cycle 8, Progression Disease
  Response rate, Tumor shrinkage rate, Liver resection rate, R0 liver resection rate( pathologically confirmed ), Progression-free survival(CT/MRI image assessed by the attending physician), Time to treatment-failure, Overall survival, Incidence of adverse events (drag-related, surgery-related) , Exploratory endpoints
Progression-free survival among the RAS wild type subpopulation | assessed every 8 weeks, up to 4 years
Exploratory analysis of the relevance of tumor size and expression level of angiogenesis-related growth factors in plasma | Baseline, Cycle 8, Progression Disease

CONTACTS AND LOCATIONS:
Overall Officials: Ichinosuke Hyodo, MD, PhD, Principal Investigator — Graduate School of Comprehensive Human Sciences, Tsukuba University, Department of Gastroenterology; Yoshihiro Kakeji, MD, PhD, FACS, Principal Investigator — Kobe University Graduate School of Medicine, Division of Gastrointestinal Surgery, Department of Surgery
Locations (1):
- EPS Corporation, Shinjuku-ku, Tokyo, Japan